CLINICAL TRIAL: NCT05035069
Title: A Randomized, Single-Blinded, Parallel Single-Center Clinical Study Exploring the Efficacy and Safety of Ciprofol and Propofol for Nonintubated General Anesthesia in Patient Undergoing Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: Efficacy and Safety of Ciprofol Compared to Propofol for Nonintubated General Anesthesia in Patients Undergoing TAVR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK3486-IIT-02
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol (Experimental)
  Interventions: Drug: Ciprofol
- Propofol (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — Ciprofol infusion, starting with 0.8 ~ 1mg/kg/h until BIS value below 60 (including 60), and then 0.2 ~ 0.6mg/kg/h until the end of the operation, ciprofol infusion was adjusted to keep the BIS value between 40-60.
  Arms: Ciprofol
Drug: Propofol — Propofol infusion, starting with 4 ~ 5mg/kg/h until BIS value below 60 (including 60), and then 1 ~ 3mg/kg/h until the end of the operation, propofol infusion was adjusted to keep the BIS value between 40-60.
  Arms: Propofol

SUMMARY:
The purpose of this study is to explore the efficacy and safety of ciprofol compared to propofol for non-intubated general anesthesia in patients undergoing transcatheter aortic valve replacement (TAVR).

DETAILED DESCRIPTION:
This is a study in subjects undergoing transcatheter aortic valve replacement (TAVR). As designed, the study will include 1-day screening period, 1-day observation period, and 1-day safety follow-up. Participants will be randomly assigned to either experimental or control group with a 1:1 allocation, with 12 subjects in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for TAVR through femoral artery access
* 1h ≤ Expected duration of surgery ≤ 3h
* Planned for general anesthesia without intubation
* 18 ≤ BMI ≤ 30
* ASA category Ⅱ～Ⅳ

Exclusion Criteria:

* Contraindications to anesthesia/sedation or a history of adverse reaction to anesthesia/sedation
* Known allergies to eggs, soy products, opioids and their antidotes, propofol, etc; Contraindications of propofol, opioids and their antidotes
* Shock and hypotension difficult that is to be corrected by vasoactive drugs in the screening period
* Hemoglobin (HB) < 10.0 g / dl (100 g / L)
* Judged by the investigator to have any other factors that make the subject unsuitable for participation in the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-09-03 (Estimated); Primary Completion 2022-02-03 (Estimated); Study Completion 2022-02-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of time that BIS value is maintained between 40 and 60 (including boundary value) | Day 1

SECONDARY OUTCOMES:
Time from the start of drug infusion to the first BIS reduction to 60 | Day 1
Time from the end of drug infusion to the recovery of BIS to 90 | Day 1
Percentage of subjects received rescue treatment | Day 1
Incidence of hypotension | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, M.D., Principal Investigator — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No